CLINICAL TRIAL: NCT02864641
Title: Mobile Technology and Online Tools to Track Adherence in Chronic Illness Patients
Acronym: OMMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 3-C Institute for Social Development (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2R44DP003101 CKD; 2R44DP003101 (NIH)
Record Dates: First submitted 2016-08-01; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Renal Insufficiency, Chronic
Keywords: chronic kidney disease; adolescents; renal disease; CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TX Group: Planet K Treatment (Experimental): Participants in the TX Group will receive access to Planet K. Families participating in the TX condition will be asked to attend a one-hour orientation session, during which study expectations and tasks will be explained. Families will be asked to watch a short 2-minute study overview video that summarizes study requirements and expectations. Parents and their children will then have the opportunity to provide informed consent/assent prior to their participation in the study. Adolescent and young adult participants will then receive a mobile phone preloaded with the Planet K app and a brief orientation to the app and associated website.
  Interventions: Behavioral: Planet K
- CO Group: Treatment-as-usual (No Intervention): A national sample of CKD participants will be recruited. Because of the inability to meet with remotely located participants for orientation and distribution of phones, these participants will be assigned to the treatment-as-usual, online control (CO) condition. For recruitment of the online control group, youth and parents interested in participating will be asked to complete a brief eligibility survey. Participants in the treatment-as-usual CO condition will not receive access to the Planet K app and website but will receive email reminders to complete surveys online at each time point.

INTERVENTIONS:
Behavioral: Planet K — Planet K is a mobile and web-based technology infrastructure specifically designed to (a) enhance youths' chronic kidney disease- and treatment-related knowledge through interactive and game-based educational materials; (b) support adherence to the treatment regimen through customized task prompts via mobile and web-based delivery; and (c) promote patient-provider communication through real-world data collection and feedback loops.
  Arms: TX Group: Planet K Treatment

SUMMARY:
The purpose of this project is to test the efficacy of Planet K, a mobile and web-based technology infrastructure specifically designed to (a) enhance youths' chronic kidney disease- and treatment-related knowledge through interactive and game-based educational materials; (b) support adherence to the treatment regimen through customized task prompts via mobile and web-based delivery; and (c) promote patient-provider communication through real-world data collection and feedback loops. Investigators will examine the effectiveness of the Planet K mobile app and website in improving treatment adherence, disease-related knowledge, transition readiness, condition management, and the psychological correlates of these variables in adolescents and young adults with chronic kidney disease (CKD).

DETAILED DESCRIPTION:
Advances in medical treatment options over the past several decades have translated into substantially higher survival rates for those who suffer with chronic illness. Consequently, the prevalence of chronic illness has risen significantly in recent years, such that one out of every four youth in the United States currently lives with a chronic illness. The health and well-being of these youth is directly impacted by the degree to which they adhere to their treatment regimen. However, treatment regimens for chronic illness can be highly complex, making adherence problematic, particularly when combined with deficits in memory and executive functioning concomitant with many chronic illnesses. Adherence also tends to deteriorate over time; the youth's motivation or commitment to treatment may decline as symptoms improve or negative side effects occur. With low adherence comes worsening symptoms and significantly greater risk for serious medical complications and mortality in young adulthood. The costs associated with low adherence, such as the need for additional care, are also substantial both for the patient and society.

While a number of factors have been found to impact treatment adherence, risk for non-adherence-across varied forms of chronic illness-is markedly elevated when the youth lacks disease- and treatment-related knowledge and when parents provide little supervision for carrying out regimen tasks. With nearly 90% of youth with chronic illness expected to survive and therefore transition from pediatric care into adult-focused healthcare systems, it is critically important to empower youth to take ownership of their own healthcare. To do so, tools there is a need to provide accessible, affordable tools that can effectively increase patients' skills and knowledge for managing their illness and support on-going adherence to their treatment regimen.

The purpose of this project is to test the efficacy of Planet K, a mobile and web-based technology infrastructure specifically designed to (a) enhance youths' chronic kidney disease- and treatment-related knowledge through interactive and game-based educational materials; (b) support adherence to the treatment regimen through customized task prompts via mobile and web-based delivery; and (c) promote patient-provider communication through real-world data collection and feedback loops. Investigators will examine the effectiveness of the Planet K mobile app and website in improving treatment adherence, disease-related knowledge, transition readiness, condition management, and the psychological correlates of these variables in adolescents and young adults with chronic kidney disease (CKD).

All participants will complete study measures at pre- and post-assessment time points. In total, participants will take part in this study for approximately 2 months from pre- to post-assessment. Families will be recruited to participate in either the treatment condition or the control group. Families in the treatment condition will receive the Planet K app and access to the associated website for the full duration of the study (4 months) between pre-test and post-test. Families in the control group will not receive access to the app and website but instead will be asked to complete a series of online questionnaires at each of the two data collection time points (pre-test, post-test).

Investigators hypothesize that greater use (i.e., dosage) and prolonged use of Planet K will: increase disease-related knowledge, treatment adherence, self-efficacy for management of CKD, current CKD self-management behaviors, perceived severity of CKD, readiness to transition to independent self-care, and perceived benefits of CKD treatment, while also decreasing perceived barriers to CKD treatment. Moreover, investigators believe that improvement of these outcomes through use of Planet K will result in more positive mental health outcomes for participants, including lower depression and higher reported quality of life. Investigators expect that those in the treatment condition will have better outcomes than those in the control group on all of these measures at both midpoint and post-assessment time points. Finally, investigators expect all participants to report high usability, quality, and value of the Planet K mobile app and website and to positively rate their experience with Planet K.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Kidney Disease diagnosis

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Knowledge of CKD | Collected at two time points: pre-test and 2 months later at study completion to measure change
  Both parents and adolescent participants will complete a consultant-created 25 item questionnaire to assess their knowledge of CKD.
End Stage Renal Disease-Adherence Questionnaire (ESRD-AQ) | Collected at two time points: pre-test and 2 months later at study completion to measure change
  Both adolescent and parent participants will complete a modified version of the End Stage Renal Disease-Adherence Questionnaire (ESRD-AQ; Kim, Y., Evangelista, L.S., Phillips, L.R., Pavlish, C., & Kopple, J.D., 2010). This 28-item measure assesses the extent to which youth adhere to the treatment plan put forth by their healthcare provider, including regular visits to the doctor, taking medications as prescribed, and following dietary recommendations. The parent version contains 22 items and the youth version contains 25 items.
Perceived Treatment Benefits | Collected at two time points: pre-test and 2 months later at study completion to measure change
  Both adolescents and their parents will report on their perceptions of the benefits and barriers of adherence to the condition treatment regimen. This measure was adapted from the Beliefs about Dietary Compliance scale (BDCS; Bennett et al, 2001) and contains 9 items on both the parent and youth versions.
STARx Transition Readiness Questionnaire | Collected at two time points: pre-test and 2 months later at study completion to measure change
  This 18-item measure assesses the extent to which youth are ready to transition to independent care and manage their health-related needs independently. Items assess adolescents' independence in scheduling doctor's appointments, remembering to take medication, finding answers to health-related questions, knowledge of their condition, and how easy/difficult these tasks are for the youth.

SECONDARY OUTCOMES:
Chronic Kidney Disease Self-Efficacy Instrument | Collected at two time points: pre-test and 2 months later at study completion to measure change
  Adolescents will complete the 25-item Chronic Kidney Disease Self-Efficacy Instrument (CKD-SE; Lin, C., Wu, C., Anderson, R., et al., 2012). This measure assesses patients' self-confidence in managing their condition, including self-confidence in (a) managing the disease autonomously, (b) integrating treatment requirements to fit new situations or social activities, (c) finding solutions to CKD-related problems, and (d) finding social support when needing help.
Self-Management:Self-Efficacy for Managing Chronic Disease Scale | Collected at two time points: pre-test and 2 months later at study completion to measure change
  Self-Efficacy for Managing Chronic Disease scale (Ritter & Lorig, 2015), a 6-item measure assessing confidence in self-management ability.
Self-Management: Partners in Health Scale | Collected at two time points: pre-test and 2 months later at study completion to measure change
  Partners in Health scale (Cordova et al. 2013), an eleven item measure assessing ability to observe and manage symptoms.
Quality of Life | Collected at two time points: pre-test and 2 months later at study completion to measure change
  Adolescents will complete a subset of 19 items from the Kidney Disease and Quality of Life-Short Form (KDQOL-SF; Hays et al., 1997). Items were modified to be more general and applicable to any medical condition. These items comprise subscales that assess patients' symptoms, burden of condition in interfering with life, cognitive functioning, social support, and difficulty sleeping.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Livet, PhD, Principal Investigator — 3-C Institute for Social Development; Janey McMillen, PhD, Principal Investigator — 3-C Institute for Social Development
Locations (1):
- 3-C Institute for Social Development, Durham, North Carolina, United States